CLINICAL TRIAL: NCT00516256
Title: CHESS: Human and Computer Mentors for Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2007-0254; 1R01CA114539-01A2 (NIH)
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Quality of Life; Cancer Information Mentor; CHESS; the Comprehensive Health Enhancement Support System; Social support; Skill-building tools
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHESS System (Experimental): CHESS System - Internet-based computer program for 6 months.
  Interventions: Behavioral: CHESS System
- Cancer Information Mentor (Experimental): Cancer Information Mentor - Phone calls to the patient for 6 months.
  Interventions: Behavioral: Cancer Information Mentor
- CHESS System + Cancer Information Mentor (Experimental): CHESS System + Cancer Information Mentor
  Interventions: Behavioral: CHESS System; Behavioral: Cancer Information Mentor

INTERVENTIONS:
Behavioral: CHESS System — Internet-based computer program for 6 months.
  Other Names: Comprehensive Health Enhancement Support System
  Arms: CHESS System; CHESS System + Cancer Information Mentor
Behavioral: Cancer Information Mentor — Phone calls to the patient for 6 months.
  Arms: CHESS System + Cancer Information Mentor; Cancer Information Mentor

SUMMARY:
The aims include:

1. To measure the effect of the three study conditions on Quality of Life (QOL).

   * CHESS and Cancer Information Mentor will not differ initially (6 weeks) or late in treatment (6 months) in QOL
   * CHESS +Cancer Information Mentor will have the largest impact on QOL (initially and late in treatment) and will be significantly better than either CHESS or Cancer Information Mentor alone.
2. To measure potential intervening or mediating processes, so that we can determine how CHESS and the Cancer Information Mentor produce associated QOL benefits.
3. To conduct exploratory use analyses examining which types of CHESS content, sequential patterns of content use, or other characteristics of use behavior are associated with greater pretest-posttest improvements in QOL.
4. To conduct a secondary analysis exploring whether men whose partners have actively used CHESS do better than those whose partners did not use CHESS.

DETAILED DESCRIPTION:
CHESS and Cancer Information Mentoring:

Researchers want to learn the best way to improve a man with prostate cancer's knowledge, coping skills, and satisfaction with decision-making and overall quality of life. This study will do this by comparing the following 3 methods of receiving information, social support, and skill training: using the CHESS system for 6 months, talking to a Cancer Information Mentor for 6 months, or using the CHESS system and talking to a Cancer Information Mentor for 6 months.

CHESS is an interactive, internet-based computer program that will provide information, social support, and skill-building techniques. CHESS provides the latest medical, social, and legal information about prostate cancer (such as information on symptoms and treatments). It also provides help in deciding what treatment to choose, advice on where participants can go for help, information on how participants can make the best use of health and human services, and a way for participants to share concerns with cancer information specialists and other survivors of prostate cancer. Participants who take part in the CHESS interactive services will not need to give their names. Participants can talk with other people by sending anonymous (your identity will be unknown) messages through the CHESS computer network.

Cancer Information Mentoring is provided by a person called a "cancer information mentor" that will give quality prostate cancer information and explain medical information and procedures. The cancer information mentor is a certified information specialist trained by the National Cancer Institute (NCI). This mentor will not provide medical advice or mental health counseling.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 3 groups. No matter which group you are assigned to, you will be loaned a computer with internet access to use in your own home (unless you have your own computer and would prefer to use it). The computer will be sent to your home, and you will be trained on how to use the computer and the CHESS system.

Participants in Group 1 will have access to the CHESS system. Participants in Group 2 will talk with a cancer information mentor. Participants in Group 3 will have access to the CHESS system and talk with a cancer information mentor.

Study Participation:

CHESS Participants in Group 1 and Group 3 who receive the CHESS internet-based program will have access to information, social support, and skill-building services. The CHESS system will keep a record of how often and for how long each part of CHESS is used. Information will also be gathered about anything you communicate in the CHESS interactions. This information will be used to figure out which parts of CHESS may be most useful. You will be provided a free 1-800 phone number for computer support if you need any help.

Cancer Information Mentoring:

Patients in Group 2 and Group 3 will have access to a cancer information mentor. The mentor will make regular telephone calls to the patient during the study. He will receive 10 calls in total (4 calls the first month, 2 calls the second month, and one call each in Months 3-6). Patients can also call the cancer information mentor whenever they wish during this period. Each call will last as long as the patient needs it to.

For patients in Group 3, the cancer information mentor will communicate with them through CHESS as well as by telephone.

Surveys:

All participants will fill out 5 surveys during this study. The surveys will include questions about health, treatment decisions, knowledge of prostate cancer, and quality of life. You will complete the first survey before you get the computer and again at 2 weeks, 6 weeks, 3 months, and 6 months after getting the computer. The surveys should take about 30 minutes to finish each time.

Length of Study:

This study will last up to a little over 6 months (about 24 weeks).

Up to 327 men and 327 support persons will take part in this multicenter study. Up to 127 participants and 127 support persons will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Being within 9 weeks of a primary diagnosis of Stage 1 or Stage 2 prostate cancer
2. Being 18 years of age or older
3. Being able to read and write English at the 6th grade level (as shown by an ability to understand the informed consent)

Exclusion Criteria:

1. Being under 18 years of age.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2007-07-03 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Effect of three study conditions on Quality of Life | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Carmack Taylor, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Hartford Hospital, Hartford, Connecticut
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org